CLINICAL TRIAL: NCT00220753
Title: Air Cleaners for Children and Adolescents With Asthma and Dog Allergy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Innlandet HF (Other)
Collaborators: Incen AG (Industry)
Responsible Party: Leif Bjarte Rolfsjord/ seksjonsoverlege, Sykehuset Innlandet HF
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AIR CLEANER TRIAL 2 SIHF; PARTIAL SPONSOR INCEN AG
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2009-07-23 (Estimated); Status verified 2009-07

CONDITIONS: Asthma; Allergy
Keywords: Dog allergy; Pet allergy; Air cleaners; HEPA filters; Air filtration; Can f1; Asthma; Children; Adolescents; Indoor environment; Indoor allergy; Perennial allergy
MeSH Terms: conditions — Asthma; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active air cleaner (Active Comparator): Two Icleen IQAir air cleaners with active filters supplied
  Interventions: Device: IQAir Allergen 100 Air cleaners
- Placebo air cleaner (Placebo Comparator): Two Icleen IQAir air cleaners with placebo filters supplied
  Interventions: Device: IQAir Allergen 100 Air cleaners

INTERVENTIONS:
Device: IQAir Allergen 100 Air cleaners — Two air cleaners are installed in the patient's room, one in his bedroom, and one in the living room. The cleaners can be run at 5 different speeds: Speed 1 filtrates 60m3 of air per hour, speed 2 filtrates 90 m3 per hour, speed 3 filtrates 130 m3 per hour, speed 4 filtrates 240 m3 per hour, and speed 5 filtrates 380 m3 per hour. A timer-on period can be pre-set for every day of the week, but the cleaner can be run even in the timer-off period, at a speed pre-set and different from the timer-on period. Different timer-on off periods cannot be selected for different days, but the different days of the week can be pre-set to apply timer-on periods or not.
  Other Names: Health Pro

SUMMARY:
The purpose is to find out if Icleen IQAir, HEPA-filter air cleaners with high capacity and pre-set speed functions, have a beneficial effect on patients with asthma and allergy to dogs.

Air cleaners will be installed in the bedrooms and living rooms in the homes of children and adolescents aged 8-17 years at the study entry, with allergy to dogs, but not to house dust mites.

The investigators will look upon the significance of this study, and of a previous study with a similar design and the same main parameters to find out if this trial supports the results of the first trial by the same project leader, or makes it likely that the seemingly beneficial effects of the first study occurred by chance.

Main parameters:

* hyperventilation cold air challenge test

Supportive parameters:

* serum ECP
* symptom scores

The trial will be a parallel, double blind placebo controlled one.

DETAILED DESCRIPTION:
Project leader: Leif Bjarte Rolfsjord, M.D., section leader, Paediatric Department Sykehuset Innlandet HF Elverum-Hamar; Ragnhild Halvorsen, M.D. Ph.D., Voksentoppen, Paediatric Clinic, Rikshospitalet; Leiv Sandvik, Ph.D. professor, research leader statistics, Competence Centre for Clinical Research, Ullevaal University Hospital

AIM:

To examine if powerful air cleaners with HEPA-filters and a pre-set speed function making it possible to run the air cleaners at a high, but noisy speed at acceptable times, and , if wanted, at a lower, but less noisy speed at other times, (Icleen IQAir®) , have a favourable effect on asthma in children and adolescents aged 8-17 years, who are allergic to dogs, but not to house dust mite. To look at this study separately, but also look upon the total results of this study and a previous study performed by the project leader.

BACKGROUND:

The first study is not yet published. We found signs of clinically significant effects of active air cleaners by the parameters ECP in serum and bronchial hyperreactivity by a cold air hyperventilation test, but the results gave p-values at the border of statistical significance, p=0.104 for FEV1 reduction, and significant results, p=0.018 for differences in the change of ECP. The number of patients included in the study was 49, a lower number than wanted in the first place. We did not find significant effects on Liz Juniper's Life Quality Scale scores. Yet, there are reasons to believe that the results of the first study may have clinical significance. A cold air hyperventilation test reflects a real life situation in interior parts of Norway, resembling outdoor winter conditions strongly. In the first study Allergy Control encasing over pillows, eiderdowns and mattresses were applied compared to placebo, but no signs of effects were found on these children aged 7 to 17 with allergy to dog or cat, but not to house dust mites. The reason to exclude house dust mite allergic patients in the first trial was to examine if encasings could have any effect on patients without house dust mite allergy, and the fact that house dust mite allergy is less common in Northern interior areas, where the trial took place. Other studies indicate, however, that air cleaners can reduce allergens from dogs and cats, but not most other indoor allergens (3). We want to perform a new trial, and publish the results from each trial in one publication, but also look upon the results of a meta-analysis of both studies. Our hope is that the two trials can give more reliable information about the effects of the air cleaners. This time, no dust analyses will be taken, because dust analyses from the first trial, sent to dr. Susanne Lau at the Charité-Virchow Clinic in Berlin, showed that the air cleaners removed considerable amounts of dust (personal message from dr. Lau). The results have been summarised in an article by Groth C et al. in Allergy in 2002, and a manuscript for an article is now sent to Allergy for publication. The efficiency of IQAir air cleaners has also been documented by Stiftung Warentest in Germany. Due to limited resources and the signs of low sensitivity in such a trial, Liz Juniper's Life Quality Scale will not be applied this time. For economic reasons, hair samples for nicotine analysis will not be taken this time.

Since the first trial was completed, an important improvement of the air cleaners has arisen. A new panel makes it possible to pre-set the air cleaners at different speeds or on and off at different times of the day, at different days of the week. Once a day, the speed can be changed to another speed or turned off, and once a day, it can be turned back to the original speed in advance. In addition, the pre-set function can be overridden manually at any time. In the first trial, the timer on and off function could turn the air cleaners off once a day and on once a day, with no active cleaning during the timer off intervals, and no weekday differentiation of the timer. This improvement increases the likelihood that the air cleaners will be used at higher (and more noisy) speeds at times when nobody is at home, resulting in lower levels of flying allergen dust levels even at times when people are at home.

In the first trial, we did not find significantly stronger effects in homes with animals than in homes without animals. Only a fourth of the homes had animals through the whole trial period. For this reason, we will only include homes without pets this time, in order to get a more homogenous population. In the first trial, we had a lower age limit of 7. This time, the lower age limit is 8, to make it easier for patients to co-operate, avoiding frustration for seven-year-olds who may be excluded due to co-operation difficulties. The reason that we require dog allergy this time, not dog or cat allergy as in the first trial, is that one trial indicates that air cleaners only reduce the amount of airborne cat allergens marginally if no cat is in the room. This trial was performed in homes with cats (5). On the other hand, a trial of effects of air cleaners in homes with dogs showed a significant reduction of dog allergens even in rooms where dogs were not present (1). The studies are difficult to compare, however, because different dust sampling methods were applied.

MATERIAL:

30 patients from Hedmark county in south-eastern Norway will be examined for the study at the start. The patients will be selected from journals of patients having visited the hospital for asthma during the previous three years, having had verified allergy against dog, but not house dust mite.

TRIAL DESIGN:

1. Active group: IQAir® air cleaners, one in the patient's bedroom, and one in the room mostly used by the patient outside the bedroom; with real pre- and main filters.
2. Placebo group: As above, but the main filter substituted by a placebo filter. If the parents of the child do not live together, and the child visits the other parent at least every second weekend, both parents will be supplied with air cleaners of the same type, with equivalent placing of the cleaners.

The air cleaners are labelled either A or B, indicating if they are real or fake. Until closing of the trial, only the manufacturer will know the code. The patients will be randomised either to A or B, with no stratification. The air cleaners are sealed. Hence, it is not possible to open them to see what kind of filters they have, without breaking the seal. Even the placebo filters will seem real, for people not accustomed to looking inside air cleaners.

Protocol attachments:

Skin prick tests and specific IgE will only be performed at visit 1. Other examinations and questions applied at both visits.

ATTACHMENT 1: Clinical examination

Height, weight, inspection of thorax, any stridor must be recorded, respiration frequency, lung auscultation. The signs recorded after the Kjell Aas scale from P0 to P6:

P0: Normal. P1: No discomfort. Slightly weakened auscultatory ventilation sound. P2: No discomfort. A few sibili (fine wheezing sounds) or rhonchi at auscultation. Prolonged audible expirium. No retractions.

P3: No discomfort at rest. Abundant obstructive sounds. Slight jugular retraction, some use of auxiliary ventilation muscles. Possibly elevated shoulders.

P4: Some discomfort at rest. Abundant obstructive sounds. Fine wheezing heard without stethoscope. Jugular/intercostal retractions. Use of auxiliary ventilation muscles. Worse (P5) after cough.

P5: Considerable discomfort at rest. Abundant obstructive sounds. Wheezing expiration. Wheezing without stethoscope. Energetic use of auxiliary ventilation muscles. Possibly slight cyanosis.

P6: Alarming obstruction. Often even inspiratory obstruction. NB! Weak respiratory sounds, but retractions and use of auxiliary muscles and tachypnoea are especially alarming. Possible cyanosis.

ATTACHMENT 2: Cold air provocation test - method Material

1. Rhes-pro® cold air unit delivering cold air, with a 5.2% CO2 content, to avoid hypocapnia at hyperventilation. The apparatus must be calibrated to give a standardised temperature, -15C of the inhaled air at lip level, and 5.2% CO2.
2. Flow volume spirometer with computer.
3. Before the test, one must make sure that there is enough air and CO2 for the unit.

Medication

Drugs that can affect the results must be avoided at a certain interval. In our study, the following drugs are withheld at the indicated intervals before the test:

* Short acting beta-2-agonist: 12 hours
* Long acting beta-2-agonist: 24 hours.
* Beta-2-agonist slow release oral drugs: Generally not used in our clinic. If yet taken : 3 days
* Theophylline slow release oral drugs: Generally not used in our clinic. If yet taken: 3 days
* Antihistamines: 7 days
* Leukotriene antagonists: 48 hours.
* Atropine derivatives (ipratropium bromide): 8 hours. After the test, the patient can be given the rest of his ordinary morning drugs.

Time of the day

1. The test should be performed at the same time every time, preferably in the morning.
2. The patient should rest for 15 minutes before the test, to avoid influence by physical exercise (bicycling, running up stairs etc.).

Test method

1. Tests performed on Mondays must be avoided to prevent influence by casual contacts and activities in the course of the weekend before the test.
2. Travels including staying overnight away from the home for more than a week should be registered, and the test should be performed more than one week after arriving home from holiday.
3. The patient must have normal clinical signs (P0) before the cold air provocation, or the test must be postponed.
4. Take flow volume test, best FEV1 out of 3 attempts. A printout of the best spirometry attempt must be stored in the research archive. The flow volume tests shall be performed in a sitting position. The patient must use a nose clip during spirometry and cold air provocation.
5. Provided FEV1 is >70% of predicted, the test is started. If <70%, it is postponed.
6. The air mixture flow is calculated by the pre-provocation best FEV1 value, by multiplying FEV1 by 20 for children less than 13 years of age at the first visit, and by 26 for the adolescents more than 13 years of age at the first visit. The patient remains sitting during the cold air provocation.
7. The patient is instructed to breathe rapidly and deeply through the mouthpiece during the provocation, which lasts for 4 minutes. In practice, the test is performed by letting the child breathe sufficiently to keep a connected balloon or ventilation bag halfway filled.
8. Spirometry with FEV1 must be performed straight before and 2 minutes after provocation.
9. MEF50 (=FEF50) at each spirometry being recorded as the spirometry giving the best FEV1 will be registered.
10. Auscultation signs immediately before each series of three spirometry attempts, and possible cough, will be registered.
11. After the post-provocation spirometry (two minutes after the provocation), salbutamol, Ventolin 0,1mg meter dose inhaler by Volumatic will be given for reversibility test; 2 puffs for patients weighing less than 45 kg, and 4 puffs for patients weighing 45 kg and more; one puff at a time; 5 inhalations per puff. New spirometry will be performed 5 minutes after giving Ventolin, and FEV1 is registered again, in absolute value, and percentage of the first value, before cold air provocation.
12. Even if the risk for acute severe asthmatic symptoms is low, a nebuliser for giving salbutamol and adrenaline for subcutaneous injection and equipment for intravenous administration of antiasthmatic drugs will be easily available.(The treatment scheme from the Norwegian Paediatric Association's acute therapy book will be applied.) Evaluation of the test results Percentage fall in FEV1 and FEF50 will be applied as a parameter of bronchial reactivity. More than 10% fall in FEV1 after cold air or more than 10% rise in FEV1 after inhalation of Ventolin, is considered significant.

Printouts of the spirometry results will be saved. Patient registration sheet cold air hyperventilation test (Printouts from spirometry to be attached).

The following data will be noted:

Time of day, hours, minute. Height (cm) Weight (kg) Assisted by (nurse) Assisted by (doctor).

Questions to be asked:

Staying away from home for more than 2 weeks last month or during trial? Staying overnight away from home last week? Staying overnight for more than a week, less than one week ago? Inhaled drugs - Ventolin, Serevent, Flutide, doses, numbers of hours ago. Other drugs, route Dose x times a day Last dose, number of hours ago

To be recorded from spirometry:

Best FEV1 (pre-test) litres per minute Temperature at mouthpiece: (will be held at -15 °C). Air flow in cold unit (litres per minute) CO2 flow in cold unit (litres per minute) Number of minutes of provocation Number of pauses Patient's performance will be recorded as good, acceptable or unacceptable.

The following values and signs noted before provocation, 2 minutes after provocation and 5 minutes after Ventolin given in a spacer (Volumatic®).

FEV1, FEV1 % increase (+) or decrease (-) of pre-test MEF50 MEF50 % of first Aas score (P0-P6) Cough Other signs or symptoms If other rescue medication is given than Ventolin in Volumatic, it must be noted.

ATTACHMENT 3: Inquiry about animal contact.

1. Are there pets in the home?
2. Did you react by nose symptoms, sneezing, cough or breathing difficulties the last time you were close to a dog without having taken drugs against asthma or allergy?
3. What kind of pet do you have in the home:

   If animal removed the last half year, how many months ago? Animal now? Number of animals? Specify if you have cat, dog, rabbit, hamster, other furred pets, budgerigar, other birds, fish, other animals
4. Are you (patient) in contact with animals outside the home? How often; what kind of animal? ATTACHMENT 4: Inquiry about smoking. The staff fill in questions to patient if the patient, or anybody else in the home smokes, and if smoking in the home totals less than 10, 10-20, or more than 20 cigarettes a day.

ATTACHMENT 5: Questions about fitted carpets, humidity, vacuum cleaners, mechanical ventilation systems.

The following questions are asked by staff to parent or accompanying person (what person will be recorded).Filled in together with:

1. Do you have fitted carpets?
2. Do you have fitted carpets in the child's bedroom?
3. Do you have fitted carpets in the living room?
4. Do you have fitted carpets in other rooms?
5. Do you think that you have more than 5 cm of dew or frost on the inside of the window of the child's bedroom?
6. Is there any smell of mould in your house?
7. Where in the house is there a smell of mould?
8. Can you see mould or rotten patches in any room?
9. If yes, where can you see it?
10. What kind of vacuum cleaner do you have?
11. Is there, except for ventilation over the kitchen stove, any kind of mechanical ventilation or air filtration in the home? ATTACHMENT 6: Symptom score The patients are asked to draw a circle around one of the numbers, from 1 through 5, indicating the degree of symptoms, 1 meaning no or never, 5 meaning many times each night, severe, always, cannot breathe through my nose or cannot breathe through my nose while sitting still, respectively. For patients taking antihistamines, the nose symptoms are valid for the last 5 days. Otherwise, the questions are applicable to the last month.

Questions to patients at Visit 1 Sep./Oct.-05:

1. Do you wake up at night due to asthma?
2. How is your asthma during daytime?
3. Do you feel your asthma when you run?
4. Is your nose stuffy at night? To patients who have taken antihistaminic agents regularly for the last month this question will be asked instead: Has your nose been stuffy in daytime for the last 5 days?
5. Is your nose stuffy during daytime? To patients who have taken antihistaminic agents regularly for the last month this question will be asked instead: Has your nose been stuffy in daytime for the last 5 days? Finally, a question is asked about strong asthma attacks last 3 months. Options for answers ar no, once or several times.

ATTACHMENT 7: Medication. Prophylactic medication will be kept constant during the trial. Doubling doses of inhaled steroids for maximum two weeks during exacerbations or airway infections, or, in patients not taking inhaled steroids daily, taking inhaled steroids for maximum two weeks during exacerbations or airway infections, will be accepted. Systemic corticosteroids in the trial period will lead to exclusion.

Ongoing medication: See section about cold air challenge (attachment 2)

Pre-trial medication:

Date prescribed or "1-3" (between 1 and 3 months ago) or ">3" (more than 3 months ago) Drug name Total amount of doses prescribed Generic name Drug type (tablets, oral mixture, injection liquid etc.) Administration route Amount per dose Measured as (ml, mg etc.) Times a day in good periods Times a day in bad periods or prodromal stages Max. duration of increased dose in days Date taken away

Medication prescribed in trial period:

Date prescribed Prescribed by Drug name Total amount of doses prescribed Generic name Drug type(tablets, oral mixture, injection liquid etc.) Administration route Amount per dose Measured as (ml, mg etc.) Times a day in good periods Times a day in bad periods or prodromal stages Max. Duration of increased dose in days Date taken away ATTACHMENT 8: Skin prick tests The skin prick tests are performed with a lancet with a one mm tip (ALK). All the tests will be performed in duplicate according to the EAACI Position paper i.e. the tests will be placed in a mirror fashion on the volar aspect of the forearm. The reactions will be read after 15 minutes. The weals are to be circumscribed by a fine filter pen or ballpoint pen on the red skin around the weal, near the weal edge. A transparent tape strip is to be pressed over the circumscription and transferred over to the registration sheet. The weal size is to be recorded by assessment of the average weal diameter. Weals with an average diameter >3 mm will be considered positive.

Skin prick test protocol - allergen extract solutions and reference solutions Skin prick tests shall be performed at the inclusion of the patients at visit 1, Sep./Oct.-05. Soluprick® extract solutions from ALK will be applied.

Specifications:

1. Birch: Soluprick® SQ "ALK Abello" (108) Silver birch 10 HEP
2. Timothy: Soluprick® SQ "ALK Abello" (225) Timothy grass 10 HEP
3. Mugwort: Soluprick® SQ "ALK Abello" (312) Mugwort 10 HEP
4. House dust mite: Soluprick® SQ "ALK Abello" (504) D. Farinae 10 HEP
5. House dust mite: Soluprick® SQ "ALK Abello" (503) D. Pteronyssin. 10 HEP
6. Mould: Soluprick® SQ "ALK Abello" (417) Cladosporium herbarum 1:20 w/v
7. Mould: Soluprick® SQ "ALK Abello" (402) Alternaria alternata 1:20 w/v
8. Dog: Soluprick® SQ "ALK Abello" (553) Dog hair 10 HEP
9. Cat: Soluprick® SQ "ALK Abello" (555) Cat hair 10 HEP
10. Horse: Soluprick® SQ "ALK Abello" (552) Horse hair 10 HEP Soluprick® "ALK Abello" Negative Control will be used as negative control, and Soluprick® "ALK Abello" Positive Control, histamine dihydrochloride 10 mg/ml (ALK) as positive control.

ATTACHMENT 9 - SPECIFIC IGE A blood sample is to be taken at visit 1 in Sep/Oct.-05, for specific IgE for the same allergens as the skin prick tests, except for D.pteronyssinus. Reagents from Pharmacia Diagnostics will be applied, and their procedures for blood sampling and analyses will be applied. EMLA "Astra-Zeneca" cream can be used if wanted as a topic anaesthetic agent before blood sampling.

ATTACHMENT 10 - serum ECP At both visits, blood samples will be taken for serum ECP. Reagents from Pharmacia Diagnostics will be used, and their manuals for blood sampling and analyses applied.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents between 8 and 17 years of age at the start of the trial (born after 01 March '88, but before 01 September '97).
* Bronchial asthma, diagnosed by a physician, and confirmed by a physician at a paediatric department of a Norwegian Hospital.
* Allergy against dogs, confirmed by skin prick test. Average infiltrate at least 4 millimetres against dog, diagnosed by a new skin prick test at entry. For details about skin prick test, see attachment no. 6.
* Having had nose or breathing symptoms by contact with dogs, when no drugs against asthma or allergy have been taken.
* Able to co-operate at cold air hyperventilation test and spirometry (see attachment no. 2).
* Given written consent (by parents of children below 12; by parents and child when above 12, but below 16; by patient when above 16).

Exclusion Criteria:

* Positive house dust mite skin prick test, with a more than 3 mm infiltrate.
* Having taken oral beta-2-agonists or theophylline preparations for the last 2 weeks before trial start, or oral steroids for the last 3 months before start of the trial.
* Active smoking.
* Dogs or cats in the home.
* Staying away from the home continuously for more than 14 days in the trial period or during the last month before trial start.
* Being an in-patient in a special department or institution for asthma and allergy in the trial period or the last 3 months before the trial.
* Having another chronic disease that can influence the results of ECP or cold air hyperreactivity tests.
* Other types of mechanical ventilation or air filtration systems in the homes, except for those for kitchen stoves.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2005-09; Primary Completion 2006-02 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Bronchial hyperactivity by cold air hyperventilation | September 2005 - February 2006

SECONDARY OUTCOMES:
Serum ECP | September 2005- February 2006
Asthma symptom score | September 2005 - February 2006
Allergic rhinitis symptom score | September 2005 - February 2006

CONTACTS AND LOCATIONS:
Overall Officials: Leif B. Rolfsjord, M.D., Principal Investigator — Sykehuset Innlandet HF; Leiv Sandvik, PhD, Study Chair — Oslo Universitetssykehus Ulleval; Ragnhild Halvorsen, M.D., Ph.D., Study Chair — Oslo Universitetssykehus Rikshospitalet; Sten Dreborg, M.D., Ph.D., Study Chair — Alingsåsv. 11, S-443 35 Lerum, Sweden
Locations (1):
- Barnepoliklinikken, Sykehuset Innlandet HF, Hamar, Norway

REFERENCES:
- [Background] Green R, Simpson A, Custovic A, Faragher B, Chapman M, Woodcock A. The effect of air filtration on airborne dog allergen. Allergy. 1999 May;54(5):484-8. doi: 10.1034/j.1398-9995.1999.00029.x. PMID 10380780
- [Background] van der Heide S, van Aalderen WM, Kauffman HF, Dubois AE, de Monchy JG. Clinical effects of air cleaners in homes of asthmatic children sensitized to pet allergens. J Allergy Clin Immunol. 1999 Aug;104(2 Pt 1):447-51. doi: 10.1016/s0091-6749(99)70391-x. PMID 10452769
- [Background] Wood RA. Air filtration devices in the control of indoor allergens. Curr Allergy Asthma Rep. 2002 Sep;2(5):397-400. doi: 10.1007/s11882-002-0073-3. PMID 12165206
- [Background] McDonald E, Cook D, Newman T, Griffith L, Cox G, Guyatt G. Effect of air filtration systems on asthma: a systematic review of randomized trials. Chest. 2002 Nov;122(5):1535-42. doi: 10.1378/chest.122.5.1535. PMID 12426250
- [Background] Gore RB, Bishop S, Durrell B, Curbishley L, Woodcock A, Custovic A. Air filtration units in homes with cats: can they reduce personal exposure to cat allergen? Clin Exp Allergy. 2003 Jun;33(6):765-9. doi: 10.1046/j.1365-2222.2003.01678.x. PMID 12801310
- [Background] Simpson A, Simpson B, Custovic A, Craven M, Woodcock A. Stringent environmental control in pregnancy and early life: the long-term effects on mite, cat and dog allergen. Clin Exp Allergy. 2003 Sep;33(9):1183-9. doi: 10.1046/j.1365-2745.2003.01679.x. PMID 12956752
- [Background] Woodcock A, Lowe LA, Murray CS, Simpson BM, Pipis SD, Kissen P, Simpson A, Custovic A; NAC Manchester Asthma and Allergy Study Group. Early life environmental control: effect on symptoms, sensitization, and lung function at age 3 years. Am J Respir Crit Care Med. 2004 Aug 15;170(4):433-9. doi: 10.1164/rccm.200401-083OC. Epub 2004 May 13. PMID 15142868
- [Background] Lowe LA, Woodcock A, Murray CS, Morris J, Simpson A, Custovic A. Lung function at age 3 years: effect of pet ownership and exposure to indoor allergens. Arch Pediatr Adolesc Med. 2004 Oct;158(10):996-1001. doi: 10.1001/archpedi.158.10.996. PMID 15466689
- [Background] Arbes SJ Jr, Cohn RD, Yin M, Muilenberg ML, Friedman W, Zeldin DC. Dog allergen (Can f 1) and cat allergen (Fel d 1) in US homes: results from the National Survey of Lead and Allergens in Housing. J Allergy Clin Immunol. 2004 Jul;114(1):111-7. doi: 10.1016/j.jaci.2004.04.036. PMID 15241352